CLINICAL TRIAL: NCT04352283
Title: Does Preprocedural Ultrasound Exam of Lumbar Spine Increase the First-pass Success Rate of Epidural Space Identification Among Obese Parturients: A Randomized Controlled Open Trial
Brief Title: Does Ultrasound Increase the First-pass Success of Epidural Space Identification in Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02752-53
Record Dates: First submitted 2020-03-29; First posted 2020-04-20 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2019-03

CONDITIONS: Epidural; Anesthesia
Keywords: ultrasound; obesity; epidural analgesia; vaginal delivery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: randomized controlled open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palpation (No Intervention): Usual method to determinate needle puncture site
- Ultrasound (Experimental): Ultrasound preprocedural exam used to determinate needle puncture site
  Interventions: Device: Preprocedural ultrasound exam of lumbar spine

INTERVENTIONS:
Device: Preprocedural ultrasound exam of lumbar spine — Preprocedural ultrasound exam of lumbar spine used to determinate needle puncture site
  Arms: Ultrasound

SUMMARY:
Obesity is associated with difficulties in epidural space catheterization. The investigators want to prove that a pre-procedural ultrasound exam of lumbar spine increase the first-pass success rate of the epidural space identification among obese parturients.

DETAILED DESCRIPTION:
This study was a randomized controlled open trial with two parallel groups.

Study was conducted in only one center : the maternity of University Hospital of Caen (Normandy, France)

Written informed consent was obtained from eligible subjects after the pre-anesthetic interview in the 8th month of pregnancy.

Operators were medical interns or residents in anesthesiology. Before inclusion, they all spent an individual interview in the aim to practice ultrasound exam of lumbar spine.

Eligible subjects were full-term parturients with pre-pregnancy BMI ≥ 30 kg/m2 undergoing vaginal delivery and receiving epidural labor analgesia. Exclusion criteria were usual contraindications for neuraxial anesthesia, marked spinal deformity, previous spinal surgery and emergency context.

The study subjects were randomly assigned to palpation or ultrasound using sealed opaque envelopes containing group allocation.

Standard monitors were applied and patients were positioned sitting during landmark identification and throughout the anesthetic procedure.

In control group, needle-puncture site was determinate by the conventional technique of cutaneous palpation. Conventional palpation of the anatomical landmarks was performed and the intercristal line (Tuffier) was assumed to cross the spine at L4 spinous process or L3-L4 interspace. The skin was marked with horizontal and vertical lines at the L3-L4 and L2-L3 interspaces.

In experimental group, ultrasound exam of lumbar spine allowed to determinate the puncture site. A systematic approach described by Balki [1] was performed, using a portative ultrasound device with a 5-2 MHz curved array probe (Samsung HM70A, Samsung medical France, St-Ouen, France).

The epidural space was located using a midline approach with loss of resistance (saline solution) using and 18-gauge Tuohy needle. After successful identification of the epidural space, a 20-gauge multiorifice epidural catheter was inserted through the Tuohy needle up to 5 cm into the epidural space.The epidural analgesia protocol was PCEA (Patient Controled Epidural Analgesia) using subsequent admixture : lévo-bupivacaïne (0,625 mg/ml), sufentanil (0,02 µ/ml), clonidine (37 µg/ml).

The primary outcome was the rate of successful epidural space identification at the first needle pass (one skin puncture without redirection).

Secondary outcomes are described further.

Early procedural complications and delivery modalities (C-section, forceps) were notified.

An interview was planned 48 hours after the procedure for each parturient in the aim to assess the maternal satisfaction and detect late procedure complications.

Assuming α = 0.05 and β = 0.2 (80% power) risks and using the χ2 test, 28 patients were required in each group.

ELIGIBILITY:
Inclusion Criteria:

* Full-term parturients (≥ 37 weeks of amenorrhea)
* With pre-pregnancy BMI ≥ 30 kg/m2
* Admit for a vaginal delivery
* Receiving labour epidural analgesia

Exclusion Criteria:

* Usual contraindications for neuraxial anesthesia (thrombocytopenia, coagulopathy, uncorrected hypovolemia, infected puncture site, intracranial hypertension)
* Emergency maternal and foetal cases
* Twin pregnancy
* Marked spinal deformity ou previous spinal surgery
* Refusal to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Success of the epidural space identification at the first needle pass | Baseline up to 1 hour
  Succes rate of the epidural space identification at the first needle pass (first skin puncture and without needle redirection) for each group

SECONDARY OUTCOMES:
Success of the epidural space identification at the first skin puncture | Baseline up to 1 hour
  Success rate of the epidural space identification at the first needle pass (first skin puncture with at least one redirection) for each group
Number of skin punctures | Baseline up to 1 hour
  Number of skin punctures per parturient
Number of needle redirections | Baseline up to 1 hour
  Number of needle redirections per parturient
Number of intervertebral space punctured | Baseline up to 1 hour
  Number of intervertebral space punctured per parturient
Duration of the epidural procedure | Baseline up to 1 hour
  Duration of the epidural procedure in seconds, measured from the first skin puncture to the test dose
Early Failed of the epidural analgesia | 30 minutes after the end of the procedure
  Early Failed epidural analgesia, defined by the epidural analgesia remplacement within 30 minutes
Verbal Rating Scale | 30 minutes and 120 minutes after the epidural procedure
  Verbal Rating Scale (VRS) of pain measured after the epidural procedure : from 0 (no itch) to 10 (worst imaginable itch)
Accidental Dural puncture | Baseline up to 1 hour
  Occurence of accidental dural puncture during the epidural procedure
Post dural puncture headache | 48 hours after the epidural procedure
  Occurence of Post dural puncture headache after the epidural procedure
Quality of epidural analgesia | 48 hours after the epidural procedure
  Maternal perception of epidural analgesia quality during the labour : from 1 (very bad) to 5 (excellent)
Maternal perception of the duration of the epidural procedure | 48 hours after the epidural procedure
  Maternal perception of epidural procedure duration : from 1(very short) to 5 (very long)

CONTACTS AND LOCATIONS:
Overall Officials: Lise-Amelie ZERAJIC, MD, Principal Investigator — Anesthesiologist Intensivist Physician
Locations (1):
- University Hospital of Cote de Nacre, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Balki M. Locating the epidural space in obstetric patients-ultrasound a useful tool: continuing professional development. Can J Anaesth. 2010 Dec;57(12):1111-26. doi: 10.1007/s12630-010-9397-y. Epub 2010 Nov 11. English, French. PMID 21063818